CLINICAL TRIAL: NCT03095534
Title: Translating 3-Step Workout for Life in a Local Senior Living Community: A Feasibility Study
Brief Title: Translating 3-Step Workout for Life in a Local Senior Living Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Liu, Chiung-ju (CJ), Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1609528804
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Frail Elderly; Muscle Weakness
Keywords: Occupational Therapy; Aging in place; Activities of daily living; Community program
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Single group with pretest and posttest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3-Step Workout for Life (Experimental): Participants will exercise at the moderate intensity three times a week for 10 weeks. The total of 30 workout sessions will consist of 18 sessions of group single-joint resistance exercise, 6 sessions of one-on-one multiple-joint resistance exercise, and 6 sessions of one-on-one activities of daily living exercise. During the resistance exercise sessions, participants will use resistance tubing to strengthen major muscle groups of the upper extremity and lower extremity. During the activities of daily living exercise, participants will practice daily tasks around the home. The community fitness staff will modify the task demand to increase the physical challenge of the task to each participant, for example, increasing travel distance.
  Interventions: Behavioral: 3-Step Workout for Life

INTERVENTIONS:
Behavioral: 3-Step Workout for Life — a 10-week moderate exercise program

SUMMARY:
The study evaluates the feasibility of a staff-lead workout program, 3-Step Workout for Life, in a local senior living community. Eligible participants will complete assessments before and after the workout program.

DETAILED DESCRIPTION:
The 3-Step Workout for Life program is designed to help older adults improve muscle strength and apply the improved muscle strength to perform activities of daily living. The 10-week workout consists of single-joint resistance exercise, multiple-joint resistance exercise, and activities of daily living exercise. Participants will exercise in small groups in a community room as well as one-on-one with the fitness staff in their home. The community fitness staff will learn the 3-Step Workout for Life program from the University partner and deliver the program.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years old and above
2. Residents of the local study community
3. Communicable in English
4. Took more than 16 seconds to complete five chair stands with arms crossed at the chest.
5. Self-reported difficulty in performing one or more activities of daily living, which must include difficulty in feeding/eating, dressing, grooming/personal hygiene, bathing/showering, using the toilet, or functional mobility/transfer.

Exclusion Criteria:

1. Aged above 90 years old.
2. Unwilling to commit to the study program 3 sessions per week for 10 weeks.
3. Plan to move away from the current community in 6 months.
4. Having three or more errors on a six-item cognitive impairment screener.
5. Having any terminal illness, cardiovascular, neurological, psychiatric, orthopedic, or cognitive impairments that are contraindications to participating in an exercise program.
6. The difficulty of performing activities of daily living is due to neurological disorders (e.g., stroke, Parkinson's), orthopedic conditions (e.g, amputees), or sensory deficits (diabetic palsy, low vision).
7. Physician's recommendation of no moderate physical exercise.
8. Receiving home health rehabilitation therapy or exercise at moderate intensity for more than twice a week (last more than 20 minutes each time).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS)-the motor skill scale | 12 weeks
  To measure motor ability required to competently complete daily activities

SECONDARY OUTCOMES:
Box and Block Test | 12 weeks
  To measure motor coordination of the upper extremity
Timed Up and Go | 12 weeks
  To measure functional mobility
30-second arm curl test | 12 weeks
  To measure muscle strength of the upper extremity
30-second chair stand test | 12 weeks
  To measure muscle strength of the lower extremity
Canadian Occupational Performance Measure | 12 weeks
  To measure self-perception of performance in everyday living

OTHER OUTCOMES:
Montreal Cognitive Assessment | 12 weeks
  Global cognitive function measure
Patient Health Questionnaire (PHQ-9 ) | 12 weeks
  To measure the degree of depression
A Three-Item Scale Assessing Pain Intensity and Interference (PEG) | 12 weeks
  To measure the degree of pain and interfering with enjoyment of life and genera activities
UCLA Loneliness Scale | 12 weeks
  To measure the degree of loneliness
Pearlin Mastery Scale | 12 weeks
  To measure personal mastery

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-ju Liu, Principal Investigator — Indiana University School of Health & Rehabilitation Sciences
Locations (1):
- Indiana University (IUPUI Campus), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu CJ, Jones LY, Formyduval A RM, Clark DO. Task-Oriented Exercise to Reduce Activities of Daily Living Disability in Vulnerable Older Adults: A Feasibility Study of the 3-Step Workout for Life. J Aging Phys Act. 2016 Jul;24(3):384-92. doi: 10.1123/japa.2015-0070. Epub 2015 Nov 19. PMID 26583695